CLINICAL TRIAL: NCT02141347
Title: A Ph1 Open-Label Multicentre Study to Assess Safety, Tolerability, PK and Anti-tumor Activity of Tremelimumab /Tremelimumab With MEDI4736 in Japanese With Advanced Solid Malignancies or Tremelimumab in Japanese With Malignant Mesothelioma
Brief Title: Ph1 to Assess Safety, Tolerability of Tremelimumab/ Tremelimumab+MEDI4736 in Japanese Solid Malignancies/ Mesothelioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Other
Other Study IDs: D4880C00010
Record Dates: First submitted 2014-05-14; First posted 2014-05-19 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Part A and B: Advanced Solid Malignancies; Part C: Malignant Mesothelioma
MeSH Terms: interventions — tremelimumab; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A (Other): Dose escalation of tremelimumab mono therapy for advanced solid malignancies
  Interventions: Drug: Tremelimumab
- Part B (Other): Combination therapy of tremelimumab and MEDI4736 for advanced solid malignancies
  Interventions: Drug: Tremelimumab; Drug: MEDI4736
- Part C (Other): Fixed dose of tremelimumab for malignant mesothelioma
  Interventions: Drug: Tremelimumab

INTERVENTIONS:
Drug: Tremelimumab — Tremelimumab administered intravenously
Drug: MEDI4736 — MEDI4736 administered intravenously.
  Arms: Part B

SUMMARY:
A Phase I, Open-Label, Multicentre Study to Assess the Safety, Tolerability, PK and Preliminary Anti-tumor Activity when given as a monotherapy of Tremelimumab or Tremelimumab in combination with MEDI4736 in Japanese Patients with Advanced Solid Malignancies, and when given as a monotherapy of tremelimumab in Second- or Third-line Treatment of Japanese Subjects with Unresectable Pleural or Peritoneal Malignant Mesothelioma

DETAILED DESCRIPTION:
Primary objectives Part A: To investigate the safety and tolerability of tremelimumab when given to Japanese patients with advanced solid malignancies and define the dose(s) for further clinical evaluation.

Part B: To investigate the safety and tolerability of tremelimumab in combination with MEDI4736 when given to Japanese patients with advanced solid malignancies and to define the dose(s) for further clinical evaluation.

Part C: To investigate the safety and tolerability of tremelimumab when given to Japanese patients with unresectable pleural or peritoneal malignant mesothelioma.

ELIGIBILITY:
Part A and B:

Inclusion Criteria: 1. Japanese aged at least 20 years old at a time of enrollment. 2. Histological or cytological confirmation of a solid malignant tumor excluding lymphoma that is refractory to standard therapies or for which no standard therapies exist. 3. ECOG Performance Status 0-1 with no deterioration over the previous 2 weeks and minimum life expectancy of 12 weeks at a time of randomization. 4. At least one lesion (measurable and/or non-measurable) that can be accurately assessed at baseline by CT, MRI or plain X-ray and is suitable for repeated assessment. 5. Adequate bone marrow, hepatic, and renal function 6. Willingness to provide consent for archival biopsy samples if available.

Exclusion Criteria: 1. Received any prior treatment with monoclonal antibody against Programmed death 1 (PD1), Programmed death ligand 1 (PD-L1) and CTLA-4 (eg, ipilimumab) 2. The last dose of prior chemotherapy or radiation therapy was received less than 2 weeks prior to randomization 3 Currently receiving systemic corticosteroids or other immunosuppressive medications or has a medical condition that requires the chronic use of corticosteroids. 4. Receipt of live attenuated vaccination within 30 days of starting tremelimumab treatment 5. Active, untreated central nervous system (CNS) metastasis (subjects with brain metastases who are identified at screening 6. History of other malignancy unless the subject has been disease-free for at least 3 years. 7. Any unresolved chronic toxicity CTCAE grade ≥2 from previous anticancer therapy at the time of randomization, 8. Major surgical procedure within 30 days of starting

Part C:

Inclusion Criteria: 1. Japanese aged 20 and over at the time of consent 2. Histologically and/or cytologically confirmed pleural or peritoneal malignant mesothelioma 3. Disease not amenable to curative surgery 4. ECOG Performance status 0-1 5. Progressed after previous receipt of 1-2 prior systemic treatments for advanced disease that included a first-line pemetrexed (or anti-folate)-based regimen in combination with platinum agent. 6. Measurable disease, defined as at least 1 lesion (measurable) that can be accurately assessed at baseline by computed tomography CT or MRI and is suitable for repeated assessment. 7. Adequate bone marrow, hepatic, and renal function Exclusion Criteria: 1. Subjects who failed more than 2 prior systemic treatment regimens for advanced malignant mesothelioma 2. Received any prior mAb against CTLA-4, PD1 or PD-L1 3. History of chronic inflammatory or autoimmune disease. 4. Symptomatic, untreated CNS metastasis. 5. Any serious uncontrolled medical disorder or active infection that would impair the subject's ability to receive investigational product. 6. History of other malignancy. 7. History of diverticulitis, inflammatory bowel disease, sarcoidosis syndrome 8. Currently receiving systemic corticosteroids or other immunosuppressive medications. 9. Vaccinated with live attenuated vaccines within 30 days prior to starting tremelimumab treatment 10. Not recovered from all toxicities associated with prior cancer treatment to acceptable baseline status, or a NCI CTCAE ver.3.0 Grade of 0 or 1

Ages: 20 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-05-22 (Actual); Primary Completion 2017-01-27 (Actual); Study Completion 2017-01-27 (Actual)

PRIMARY OUTCOMES:
Adverse event | From time of informed consent to 90 days after the last dose
  To investigate the safety and tolerability of tremelimumab and/ or MEDI4736 when given to Japanese patients

CONTACTS AND LOCATIONS:
Locations (11):
- Japan (11):
  - Research Site, Bunkyō City
  - Research Site, Chūōku
  - Research Site, Hiroshima
  - Research Site, Nagoya
  - Research Site, Nishinomiya-shi
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Sunto-gun
  - Research Site, Ube-shi
  - Research Site, Yokohama

REFERENCES:
- [Derived] Fujiwara Y, Takahashi Y, Okada M, Kishimoto T, Kondo S, Fujikawa K, Hayama M, Sugeno M, Ueda S, Komuro K, Lanasa M, Nakano T. Phase I Study of Tremelimumab Monotherapy or in Combination With Durvalumab in Japanese Patients With Advanced Solid Tumors or Malignant Mesothelioma. Oncologist. 2022 Sep 2;27(9):e703-e722. doi: 10.1093/oncolo/oyac099. PMID 35671201